CLINICAL TRIAL: NCT04684368
Title: A Phase 2 Trial of Chemotherapy Followed by Response-Based Whole Ventricular &Amp; Spinal Canal Irradiation (WVSCI) for Patients With Localized Non-Germinomatous Central Nervous System Germ Cell Tumor
Brief Title: A Study of a New Way to Treat Children and Young Adults With a Brain Tumor Called NGGCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACNS2021; NCI-2020-13175 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACNS2021 (Other: Children's Oncology Group); ACNS2021 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2020-12-15; First posted 2020-12-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Central Nervous System Nongerminomatous Germ Cell Tumor; Choriocarcinoma; Embryonal Carcinoma; Immature Teratoma; Malignant Teratoma; Mixed Germ Cell Tumor; Pineal Region Germ Cell Tumor; Pineal Region Immature Teratoma; Pineal Region Yolk Sac Tumor; Suprasellar Germ Cell Tumor
MeSH Terms: conditions — Choriocarcinoma; Carcinoma, Embryonal; Teratoma | interventions — Specimen Handling; Carboplatin; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; Ifosfamide; Magnetic Resonance Spectroscopy; Mesna; pegfilgrastim; pegylated granulocyte colony-stimulating factor; Peripheral Blood Stem Cell Transplantation; Radiotherapy; Radiation; Second-Look Surgery; Reoperation; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Plan A (chemotherapy, WVSCI, second-look surgery if needed) (Experimental): See Outline in Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Etoposide; Biological: Filgrastim; Drug: Ifosfamide; Procedure: Magnetic Resonance Imaging; Drug: Mesna; Biological: Pegfilgrastim; Other: Questionnaire Administration; Radiation: Radiation Therapy; Procedure: Second-Look Surgery
- Plan B (chemotherapy, HDCSCR, second-look surgery if needed) (Experimental): See Outline in Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Etoposide; Biological: Filgrastim; Drug: Ifosfamide; Procedure: Magnetic Resonance Imaging; Drug: Mesna; Biological: Pegfilgrastim; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Questionnaire Administration; Radiation: Radiation Therapy; Procedure: Second-Look Surgery; Drug: Thiotepa

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of CSF and blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Biological: Filgrastim — Given subcutaneously (SC) or IV
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Mesna — Given IV or orally
  Other Names: 2-Mercaptoethanesulfonate, Sodium Salt; Ausobronc; D-7093; Filesna; Mercaptoethane Sulfonate; Mercaptoethanesulfonate; Mesnex; Mesnil; Mesnum; Mexan; Mistabron; Mistabronco; Mitexan; Mucofluid; Mucolene; UCB 3983; Uromitexan; Ziken
Biological: Pegfilgrastim — Given SC
  Other Names: Dulastin; Filgrastim SD-01; filgrastim-SD/01; Fulphila; Fylnetra; G-Lasta; HSP-130; Jinyouli; Neulasta; Neulastim; Neupopeg; Nyvepria; PEG-filgrastim; Pegcyte; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Nyvepria; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim Biosimilar PF-06881894; Pegfilgrastim Biosimilar Udenyca; Pegfilgrastim Biosimilar Ziextenzo; Pegfilgrastim-apgf; Pegfilgrastim-bmez; Pegfilgrastim-cbqv; Pegfilgrastim-fpgk; Pegfilgrastim-jmdb; Pegfilgrastim-pbbk; Pegylated G-CSF; Pegylated GCSF; Pegylated Granulocyte Colony Stimulating Factor; PF-06881894; SD-01; SD-01 sustained duration G-CSF; Stimufend; Tripegfilgrastim; Udenyca; Ziextenzo
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo PBSC transplant
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood; Peripheral Blood Progenitor Cell Transplantation; PERIPHERAL BLOOD STEM CELL TRANSPLANT; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
  Arms: Plan B (chemotherapy, HDCSCR, second-look surgery if needed)
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo WVSCI radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Plan A (chemotherapy, WVSCI, second-look surgery if needed)
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Plan B (chemotherapy, HDCSCR, second-look surgery if needed)
Procedure: Second-Look Surgery — Undergo second-look surgery if needed
  Other Names: Reoperation; Repeat Surgery; Second Look; Surgical Revision
Drug: Thiotepa — Given IV
  Other Names: 1,1',1''-Phosphinothioylidynetrisaziridine; Girostan; N,N', N''-Triethylenethiophosphoramide; Oncotiotepa; SH 105; SH-105; SH105; STEPA; Tepadina; Tepylute; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene Thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312
  Arms: Plan B (chemotherapy, HDCSCR, second-look surgery if needed)

SUMMARY:
This phase II trial studies the best approach to combine chemotherapy and radiation therapy (RT) based on the patient's response to induction chemotherapy in patients with non-germinomatous germ cell tumors (NGGCT) that have not spread to other parts of the brain or body (localized). This study has 2 goals: 1) optimizing radiation for patients who respond well to induction chemotherapy to diminish spinal cord relapses, 2) utilizing higher dose chemotherapy followed by conventional RT in patients who did not respond to induction chemotherapy. Chemotherapy drugs, such as carboplatin, etoposide, ifosfamide, and thiotepa, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays or high-energy protons to kill tumor cells and shrink tumors. Studies have shown that patients with newly-diagnosed localized NGGCT, whose disease responds well to chemotherapy before receiving radiation therapy, are more likely to be free of the disease for a longer time than are patients for whom the chemotherapy does not efficiently eliminate or reduce the size of the tumor. The purpose of this study is to see how well the tumors respond to induction chemotherapy to decide what treatment to give next. Some patients will be given RT to the spine and a portion of the brain. Others will be given high dose chemotherapy and a stem cell transplant before RT to the whole brain and spine. Giving treatment based on the response to induction chemotherapy may lower the side effects of radiation in some patients and adjust the therapy to a more efficient one for other patients with localized NGGCT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To monitor outcome to ensure that children and young adults with localized central nervous system (CNS) non-germinomatous germ cell tumors (NGGCT) treated with induction chemotherapy followed by response evaluation and whole ventricular + spinal canal irradiation (WVSCI) will maintain the excellent 2-year progression free survival (PFS) rate as compared to ACNS0122 (NCT00047320).

II. To improve disease control by decreasing the number of spinal relapses for patients who achieve a complete response (CR) or partial response (PR) and receive WVSCI as compared to whole ventricular radiation on ACNS1123 (NCT01602666).

SECONDARY OBJECTIVES:

I. To estimate the response rates to induction chemotherapy and WVSCI for localized NGGCT patients who achieve a CR/PR.

II. To estimate the PFS and overall survival (OS) for localized NGGCT patients who achieve a CR/PR and receive WVSCI.

III. To estimate the PFS and OS for patients with less than a CR/PR following Induction who subsequently receive high-dose chemotherapy with peripheral stem cell rescue (HDCSCR).

IV. To estimate the response rate for patients with less than a CR/PR following Induction who subsequently receive HDCSCR.

EXPLORATORY OBJECTIVES:

I. To prospectively compare outcomes based on radiation modality, photon versus proton, including cognitive, social and behavioral functioning, auditory, and neuro-endocrine function.

II. To compare spinal column growth and cell counts following radiation as measured by height and weight, and complete blood count (CBC) values during and after radiation therapy, based on treatment modality (photon versus [vs.] proton therapy) and planned inclusion/exclusion of the vertebral body in patients < 13 years of age.

III. To compare local vs. central review recommendations for second-look surgery and document barriers for performing such surgeries as well as their clinical benefit in pediatric NGGCT.

IV. To prospectively evaluate and longitudinally model the cognitive, social, and behavioral functioning of children and young adults with localized CNS NGGCT with testing as per the Children's Oncology Group (COG) Standardized Neuropsychological and Behavioral Battery.

V. To evaluate patterns of disease recurrence/failure with respect to radiation dose distribution.

OUTLINE:

INDUCTION CHEMOTHERAPY: Patients receive carboplatin intravenously (IV) over 15-60 minutes on day 1 and etoposide IV over 90-120 minutes on days 1-3 of cycles 1, 3, and 5. Patients also receive ifosfamide IV over 60 minutes and etoposide IV over 60-120 minutes on days 1-5 of cycles 2, 4, and 6. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

Patients are assigned to 1 of 2 plans (ventricular + spinal canal irradiation [WVSCI] or high-dose chemotherapy with peripheral stem cell rescue [HDCSCR]) based on response to induction chemotherapy:

* Patients who achieve radiographic CR/PR with marker normalization proceed to WVSCI. Patients who achieve radiographic CR without marker normalization proceed to HDCSCR.
* Patients who achieve less than radiographic CR/PR with marker normalization proceed to second-look surgery (unless contraindicated). If second-look surgery reveals mature teratoma or non-viable tumor, proceed to WVSCI. If second-look surgery reveals viable tumor, proceed to HDCSCR. Patients who are unable to undergo second-look surgery are removed from protocol therapy but remain on study for follow-up.
* Patients who achieve less than radiographic CR/PR without marker normalization proceed to second-look surgery (unless contraindicated). Patients then proceed to HDCSCR regardless of whether or not a second-look surgery is performed.
* Patients who achieve radiographic PR without marker normalization proceed to second-look surgery (unless contraindicated). Patients then proceed to HDCSCR regardless of whether or not a second-look surgery is performed.

PLAN A (WVSCI THERAPY): Within 6 weeks of the end of induction chemotherapy or second-look surgery, patients undergo WVSCI once daily (QD) for 5 days weekly (17 fractions followed by a boost dose for 13 fractions) for 6 weeks in the absence of disease progression or unacceptable toxicity.

PLAN B (CONSOLIDATION THERAPY [HDCSCR]): Within 6-8 weeks of the end of induction chemotherapy or second-look surgery, patients receive etoposide IV and thiotepa IV over 3 hours on days -5 to -3 and undergo peripheral blood stem cell (PBSC) transplant on day 0. Patients then undergo radiation therapy QD for 5 days weekly (20 fractions followed by a boost dose for 10 fractions) for 6 weeks in the absence of disease progression or unacceptable toxicity.

Patients also undergo magnetic resonance imaging (MRI), as well as collection of cerebral spinal fluid (CSF) and blood sample throughout the trial.

After completion of study treatment, patients are followed for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >= 3 years and < 30 years at the time of study enrollment
* Patients must be newly diagnosed with localized primary CNS NGGCT of the suprasellar and/or pineal region by pathology and/or serum or cerebrospinal fluid (CSF) elevation of AFP above institutional normal or > 10 ng/mL or human chorionic gonadotropin (hCG) beta > 100 mIU/mL as confirmed by Rapid Central Marker Screening Review on APEC14B1-CNS. Suprasellar, pineal and bifocal tumors are included. (CSF tumor markers and cytology must be within 31 days prior to enrollment and start of protocol therapy [repeat if necessary]. Serum tumor markers, AFP and hCGbeta must be within 7 days prior to enrollment and start of protocol therapy [repeat if necessary]). Basal ganglia or other primary sites are excluded
* Patients with any of the following pathological elements are eligible: endodermal sinus (yolk sac), embryonal carcinoma, choriocarcinoma, malignant/immature teratoma and mixed germ cell tumor (GCT) (i.e., may include some pure germinoma) if malignant elements listed above are present. Patients with only mature teratoma are excluded. Patients with pure germinoma admixed with mature teratoma are excluded (would be eligible for pure germinoma protocols)
* Patients must have a cranial MRI with and without gadolinium at diagnosis/prior to enrollment. If surgical resection is performed, patients must have pre-operative and post operative brain MRI with and without gadolinium. The post operative brain MRI should be obtained within 72 hours of surgery. If patient has a biopsy only, post-operative brain MRI is recommended but not required (within 31 days prior to study enrollment and start of protocol therapy )
* Patients must have a spine MRI with gadolinium obtained at diagnosis/prior to enrollment. Spine MRI with and without gadolinium is recommended (within 31 days prior to study enrollment and start of protocol therapy)
* Lumbar CSF must be obtained prior to study enrollment unless medically contraindicated. If a patient undergoes surgery and lumbar CSF cytology cannot be obtained at the time of surgery, then it should be performed at least 10 days following surgery and prior to study enrollment. False positive cytology can occur within 10 days of surgery
* Patients must have RAPID CENTRAL TUMOR MARKER REVIEW CSF tumor markers obtained prior to enrollment unless medically contraindicated. Ventricular CSF obtained at the time of CSF diversion procedure (if performed) is acceptable for tumor markers but lumbar CSF is preferred. In case CSF diversion and biopsy/surgery are combined, CSF tumor markers should be collected first
* Peripheral absolute neutrophil count (ANC) >= 1000/uL (within 7 days prior to enrollment)
* Platelet count >= 100,000/uL (transfusion independent) (within 7 days prior to enrollment)
* Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions) (within 7 days prior to enrollment)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows (within 7 days prior to enrollment):

  * Age: Maximum serum creatinine (mg/dL)

    * 3 to < 6 years: 0.8 (male), 0.8 (female)
    * 6 to < 10 years: 1 (male), 1 (female)
    * 10 to < 13 years: 1.2 (male), 1.2 (female)
    * 13 to < 16 years: 1.5 (male), 1.4 (female)
    * >= 16 years: male (1.7), 1.4 (female)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (within 7 days prior to enrollment)

  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L
* Central nervous system function defined as:

  * Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
  * Patients must not be in status epilepticus, coma or assisted ventilation prior to study enrollment
* Protocol therapy must begin within 31 calendar days of definitive surgery or clinical diagnosis, whichever is later. If a biopsy only was performed, the biopsy date will be considered the date of definitive surgery. For patients who have a biopsy or incomplete resection at diagnosis followed by additional surgery, the date of the last resection will be considered the date of definitive surgery.
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met
* NEUROCOGNITIVE FUNCTION AND QUALITY OF LIFE ASSESSMENT:
* English-, Spanish-, or French- speaking

  * Note: Patients who speak a language other than English, Spanish, or French will be allowed to participate in ACNS2021 but will not complete the neurocognitive and quality of life assessments
* No known history of neurodevelopmental disorder prior to diagnosis of NGGCT (e.g., Down syndrome, fragile X, William syndrome, intellectual disability). Patients with NF1 will be allowed to participate
* Additional eligibility criteria for the COG Standardized Neuropsychological Battery only: must be at a site that has a psychologist to administer the battery

  * Note: If not eligible for the COG Standardized Battery, patients should still complete the Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2), Pediatric Quality of Life Inventory (PedsQL), Adaptive Behavior Assessment System Third Edition (ABAS-3), and Behavior Assessment System for Children, Third Edition (BASC-3) questionnaires

Exclusion Criteria:

* Patients with tumors located outside the ventricles (i.e., basal ganglia, thalamus)
* Patients with only mature teratoma and non-elevated markers upon tumor sampling at diagnosis
* Patients who have received any prior tumor-directed therapy for their diagnosis of NGGCT other than surgical intervention and corticosteroids
* Patients with metastatic disease (i.e., MRI evaluation, lumbar CSF cytology or intraoperative evidence of dissemination)
* Female patients who are pregnant, since fetal toxicities and teratogenic effects have been noted for several of the study drugs

  * Note: Serum and urine pregnancy tests may be falsely positive due to HCGbeta-secreting germ cell tumors. Ensure the patient is not pregnant by institutional standards
* Lactating females who plan to breastfeed their infants
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation

Ages: 3 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2029-12-21 (Estimated); Study Completion 2029-12-21 (Estimated)

PRIMARY OUTCOMES:
Failure rate | Within 2 years of enrollment
  Will be measured by the number of progressions or deaths within 2 years of enrollment for the cohort treated with whole ventricular + spinal canal irradiation (WVSCI). The final analysis will include an exact binomial confidence interval of the failure rate for each of the failure types (local, distant/spinal or both) without adjustment for multiplicity.
Spinal failure rate | Within 2 years of enrollment
  Will be measured by the number of spinal relapses (spine alone or distant relapses including the spine) within 2 years of enrollment in patients treated with WVSCI. The final analysis will include an exact binomial confidence interval of spinal failure rate.

SECONDARY OUTCOMES:
Radiographic complete response (CR)/partial response (PR) with marker normalization rate post induction/second-look surgery | Approximately 6 to 9 months post-treatment initiation
  Will be assessed in patients treated with induction chemotherapy. Will be estimated using an exact binomial approach and its confidence interval.
Radiographic complete response (CR)/partial response (PR) with marker normalization rate post high-dose chemotherapy with peripheral stem cell rescue (HDCSCR) | Up to 2 years post-treatment initiation
  Will be assessed in patients treated with HDCSCR. Will be estimated using an exact binomial approach and its confidence interval.
Progression-free survival (PFS) | From enrollment until disease progression or death from any cause for patients with events, and until final follow up for those who are event free at the time of analysis, assessed up to 10 years
  Will be estimated separately for those treated with WVSCI and with HDCSCR + radiation therapy. Kaplan-Maier based PFS curve estimates will be included, where patients who are lost to follow up will be treated as censored observations as part of the primary analyses.
Overall survival (OS) | From enrollment until death from any cause for patients with events and until final follow up for those who are alive at the time of analysis, assessed up to 10 years
  Will be estimated separately for those treated with WVSCI and with HDCSCR + radiation therapy. Kaplan-Maier based OS curve estimates will be included, where patients who are lost to follow up will be treated as censored observations as part of the secondary analyses.
Patterns of disease recurrence/failure | Up to 10 years
  Will be analyzed in an exploratory manner with respect to radiation dose distribution.

OTHER OUTCOMES:
Change in intelligence scores within each treatment arm | Baseline up to 60 months post-treatment initiation
  Will be assessed by the Wechsler Preschool and Primary Scale of Intelligence 4th Edition (WPPSI-IV), Wechsler Intelligence Scale for Children 5th Edition (WISC-V), and the Wechsler Adult Intelligence Scale 4th Edition (WAIS-IV), depending on patient's age. One-sample confidence intervals will be used to estimate mean pairwise changes in intelligence scores between 2 time points within each treatment arm.
Change in intelligence scores between treatment arms | Baseline up to 60 months post-treatment initiation
  Will be assessed by the Wechsler Preschool and Primary Scale of Intelligence 4th Edition (WPPSI- IV), Wechsler Intelligence Scale for Children 5th Edition (WISC V), and the Wechsler Adult Intelligence Scale 4th Edition (WAIS-IV), depending on patient's age. A 2-sample confidence interval approach will be used to estimate the difference in score changes between the two cohorts (WVSCI versus HDCSCR) in order to describe differential effects of the 2 treatment strategies.
Change in processing speed/attention within each treatment arm | Baseline up to 60 months post-treatment initiation
  Will be assessed by the WISC-V or WAIS-IV processing speed index tasks. One-sample confidence intervals will be used to estimate mean pairwise changes in scores between 2 time points within each treatment arm.
Change in processing speed/attention between the two treatment arms | Baseline up to 60 months post-treatment initiation
  Will be assessed by the WISC-V or WAIS-IV processing speed index tasks. A 2-sample confidence interval approach will be used to estimate the difference in score changes between the two cohorts (WVSCI versus HDCSCR) in order to describe differential effects of the 2 treatment strategies.
Change in immediate visual memory within each arm | Baseline up to 60 months post-treatment initiation
  Will be assessed by the Children's Memory Scale and California Verbal Learning Test. One-sample confidence intervals will be used to estimate mean pairwise changes in scores between 2 time points within treatment arms, as appropriate.
Change in social-emotional functioning within each arm | Baseline up to 60 months post-treatment initiation
  Will be assessed by the Behavior Assessment System for Children - 3rd Edition. One-sample confidence intervals will be used to estimate mean pairwise changes in scores between 2 time points within treatment arms, as appropriate.
Change in adaptive functioning within each arm | Baseline up to 60 months post-treatment initiation
  Will be assessed by the Adaptive Behavior Assessment System - 3rd Edition. One-sample confidence intervals will be used to estimate mean pairwise changes in scores between 2 time points within treatment arms, as appropriate.
Change in health-related quality of life within each arm | Baseline up to 60 months post-treatment initiation
  Will be assessed by the Pediatric Quality of Life Inventory version 4.0. One-sample confidence intervals will be used to estimate mean pairwise changes in scores between 2 time points within treatment arms, as appropriate.
Change in health-related quality of life between the two treatment arms | Baseline up to 60 months post-treatment initiation
  Will be assessed by the Pediatric Quality of Life Inventory version 4.0. 2-sample confidence interval approach will be used to estimate the difference in score changes between the two cohorts (WVSCI versus HDCSCR) in order to describe differential effects of the 2 treatment strategies.
Radiation modality (proton versus photon) | Up to 10 years
  Will summarize and compare functional outcomes, including cognitive, social and behavioral functioning, and auditory and neuro-endocrine function, in the context of the radiation therapy modality used. Two sample t-tests for specified timepoints within each of the two treatment cohorts (WVSCI versus HDCSCR) will be used for comparisons.
Growth comparisons following radiation by radiation modality | Up to 10 years
  Will compare early and late outcomes for proton and photon therapy with and without vertebral body sparing. Height and weight of subjects who are < 13 years at the time of radiation therapy will be collected until subjects go off study or reach the age of 21, whichever is earlier. Percentile values standardizing height and weight based on appropriate growth curves will be used to compare cohorts treated with proton- versus photon-based radiation therapy.
Complete blood count values following radiation by radiation modality | Up to 1 year post treatment initiation
  Complete blood count values during radiation therapy will be used to compare these outcomes in the context of proton- versus photon-based radiation therapy.
Local versus central review recommendations for second-look surgery | Up to 1 year post treatment initiation
  Will summarize the local versus central review recommendations for second-look surgery and document any discrepancies.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M MacDonald, Principal Investigator — Children's Oncology Group
Locations (164):
- United States (147):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Cancer Care Specialists - Reno, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
- Australia (5):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (11):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Christchurch Hospital, Christchurch, New Zealand